CLINICAL TRIAL: NCT07399158
Title: CROSSROAD: A Prospective Multicenter Observational Study on the Efficacy of Treatment Regimen Switch With Re-induction Chemotherapy Versus Direct Radiotherapy in Locally Advanced Nasopharyngeal Carcinoma Patients With Inadequate Response (SD/PD) After Induction Chemotherapy
Brief Title: CROSSROAD: Treatment Regimen Switch - Re-induction Chemotherapy vs. Direct Radiotherapy in LANPC With Inadequate Response to Induction Chemotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiaojuan Guo, Director, Department of Head and Neck Radiation Oncology, Clinical Professor, Fujian Cancer Hospital
Other Study IDs: 2026-01-17
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Re-induction Chemotherapy Group: This group consists of patients with locally advanced nasopharyngeal carcinoma (LANPC) who did not achieve a sufficient response (stable disease or disease progression) after two cycles of induction chemotherapy. These patients will receive re-induction chemotherapy followed by radiotherapy as part of their treatment regimen.
- Direct Radiotherapy Group: This group consists of patients with locally advanced nasopharyngeal carcinoma (LANPC) who did not achieve a sufficient response (stable disease or disease progression) after two cycles of induction chemotherapy. These patients will receive direct radiotherapy without re-induction chemotherapy.

SUMMARY:
This study aims to compare the efficacy of two treatment strategies-re-induction chemotherapy followed by radiotherapy versus direct radiotherapy-in patients with locally advanced nasopharyngeal carcinoma (LANPC) who did not achieve a sufficient response (stable disease or disease progression) after two cycles of induction chemotherapy. The study will enroll patients who have completed two cycles of induction chemotherapy and have not achieved a partial or complete response. Participants will receive one of the two treatment options to evaluate their three-year progression-free survival (PFS) and other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 to 70 years old.

Histologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO Type II/III).

Initial treatment with no distant metastasis: Locally advanced nasopharyngeal carcinoma (according to the AJCC/UICC 9th edition staging, stage II-III, i.e., T3-4N0-3M0 or T1-2N2-3M0).

Completion of two cycles of standard induction chemotherapy (such as TPF, GP, TP, etc.).

Post-induction chemotherapy evaluation: Disease stability (SD) or disease progression (PD) after two cycles of induction chemotherapy, as assessed by RECIST 1.1 criteria, based on enhanced MRI of the nasopharynx.

ECOG Performance Status (PS): 0-1.

Bone marrow, liver, and kidney function: Sufficient to tolerate concurrent chemoradiotherapy (specific criteria to be referenced).

Informed consent: Voluntary participation in the study and signing of written informed consent.

Exclusion Criteria:

History of head and neck tumor radiotherapy or any other malignant cancer history (except for cured non-melanoma skin cancer).

Partial response (PR) or complete response (CR) after induction chemotherapy.

Severe uncontrolled comorbidities, such as unstable angina, congestive heart failure, severe chronic obstructive pulmonary disease (COPD), or uncontrolled diabetes mellitus.

Active infection or severe immunodeficiency diseases.

Pregnant or breastfeeding women.

Any mental or social disorders that may interfere with study evaluation or compliance.

Other conditions deemed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients aged 18-70 years with histologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO Type II/III) and no distant metastasis. Eligible participants must have completed two cycles of standard induction chemotherapy (e.g., TPF, GP, or TP), and the post-induction treatment evaluation must show stable disease (SD) or disease progression (PD) according to RECIST 1.1 criteria. Patients should have an ECOG Performance Status (PS) of 0-1 and adequate bone marrow, liver, and kidney function to tolerate concurrent chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Baseline, 1 year, 2 years, 3 years
  The primary endpoint of this study is to compare the 3-year progression-free survival (PFS) rate between the two treatment groups. Disease progression will be assessed using RECIST 1.1 criteria, with imaging exams (such as MRI) used to monitor tumor size and progression.

SECONDARY OUTCOMES:
Local Regional Recurrence-Free Survival | Baseline, 1 year, 2 years, 3 years
  This secondary endpoint will evaluate the 3-year local regional recurrence-free survival (LRRFS) rate between the two treatment groups.
Overall Survival | Baseline, 1 year, 2 years, 3 years
  This secondary endpoint will evaluate the 3-year overall survival (OS) rate. The OS rate will be compared between the re-induction chemotherapy followed by radiotherapy group and the direct radiotherapy group.
Distant Metastasis-Free Survival | Baseline, 1 year, 2 years, 3 years
  This secondary endpoint will evaluate the 3-year distant metastasis-free survival (DMFS) rate.
Complete Response Rate after Radiotherapy | 3 months post-treatment
  This secondary endpoint will assess the rate of complete response (CR) after radiotherapy.
3-4 Grade Acute Toxicity Incidence | through study completion, an average of 4-6 months
  This secondary endpoint will assess the incidence of grade 3 or 4 acute toxicity, based on the Common Terminology Criteria for Adverse Events (CTCAE) scale. The toxicity will be assessed during the course of the treatment.

IPD SHARING:
Plan to Share IPD: No